CLINICAL TRIAL: NCT05599672
Title: Co-Use of Opioid Medications and Alcohol Prevention Study (COAPS)
Brief Title: Co-Use of Opioid Medications and Alcohol Prevention Study
Acronym: COAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jerry Cochran, PhD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00152822; 1R34AA029447-01A1 (NIH)
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Drinking; Opioid Use
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: This study will test the Adapt/manualize an Alcohol-targeted Brief Intervention-Medication Therapy Management (ABI-MTM) intervention compared to standard medication counseling
Who Masked: Outcomes Assessor
Masking Description: The assessor is blinded to the intervention condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol-targeted Brief Intervention-Medication Therapy Management (Experimental): Alcohol-targeted Brief Intervention-Medication Therapy Management (ABI-MTM) intervention is a pharmacy-based medication management intervention, combined with Screening, Brief Intervention, and Referral to Treatment
  Interventions: Behavioral: Alcohol-targeted Brief Intervention-Medication Therapy Management
- Standard medication counseling (Active Comparator): Standard Medication Counseling (SMC) (1) will offer counseling, (2) document counseling was offered, (3) offer a counseling process for patients not present, and (4) discuss generic substitution. Following this session, in the second SMC component, participants will be emailed/mailed (according to participant preference) safety information about co-use of alcohol and opioids
  Interventions: Behavioral: Standard medication counseling

INTERVENTIONS:
Behavioral: Alcohol-targeted Brief Intervention-Medication Therapy Management — Alcohol-targeted Brief Intervention-Medication Therapy Management (ABI-MTM) intervention is a pharmacy-based medication management intervention, combined with Screening, Brief Intervention, and Referral to Treatment. ABI-MTM includes 5 core elements. A common duration for medication counseling in outpatient pharmacies a single 30-45 minute session. These include a medication review, a personal medication record, a medication action plan, a brief motivational intervention, and documentation and follow up.
  Arms: Alcohol-targeted Brief Intervention-Medication Therapy Management
Behavioral: Standard medication counseling — Standard Medication Counseling (SMC) will be the treatment as usual condition in this study and was chosen/developed following Gold et al.'s guide for selecting control conditions in behavioral intervention studies. For the first component, all SMC participants will receive a single 5-10 minute medication information/counseling session delivered by a pharmacist, other than the study pharmacist, that possesses a similar level of education and professional licensing. The content of this session follows federal and state pharmacy requirements requiring pharmacists to: (1) offer counseling, (2) document counseling was offered, (3) offer a counseling process for patients not present (not applicable to this study given all patients must screen in person), and (4) discuss generic substitution. Following this session, in the second SMC component, participants will be emailed/mailed (according to participant preference) safety information about co-use of alcohol and opioids.
  Arms: Standard medication counseling

SUMMARY:
Previous research, including that of this team, shows that a significant portion of those regularly using opioids-particularly filling opioids at community pharmacies-also are involved in the co-use of alcohol. This study proposes to adapt a previously developed intervention for opioid medication misuse; test its acceptability, feasibility, and preliminary efficacy; and identify barriers and facilitators to large-scale research and system-level implementation. Results of this study will directly inform a fully-powered subsequent multisite trial.

DETAILED DESCRIPTION:
Co-use of alcohol and opioid medications is known to be a serious health/safety hazard-yet persists despite these negative ramifications. With limited information available within peer-reviewed literature, large-scale system and clinical research have demonstrated 24-38% of those with alcohol use disorders also have an opioid addiction, with rates of past 30-day opioid medication misuse among those seeking alcohol treatment as high as 68%. Research from this group has shown that among community pharmacy patients receiving opioid medications for pain management, approximately 20-30% are engaged in co-use of alcohol. Community pharmacy is a highly valuable but underutilized resource and setting for identification and intervention to address the US opioid epidemic. The investigators propose to adapt, manualize, and test the acceptability, feasibility, and preliminary efficacy of an Alcohol-targeted Brief Intervention-Medication Therapy Management (ABI-MTM) intervention with community pharmacy patients. ABI-MTM will be a pharmacy-based medication management intervention, combined with Screening, Brief Intervention, and Referral to treatment that will target: (1) alcohol use elimination during opioid treatment OR (2) non-opioid pain management substitution (in consultation with the prescriber). The investigators will conduct a small-scale trial in 3 community pharmacy locations wherein the investigators will randomize patients with heavy alcohol use and with non-heavy alcohol use (1-to-1 ratio) to ABI-MTM (n=20) or standard medication counseling (SMC, n=20). Results will demonstrate intervention acceptability, feasibility, and preliminary efficacy. This study will also work to identify pharmacy system and practice-level barriers and facilitators for universal alcohol screening and intervention among opioid recipients. This study will also work to identify pharmacy system and practice-level barriers and facilitators for universal alcohol screening and intervention among opioid recipients. The investigators will develop a mixed methods assessment guide to interview pharmacy technicians (N=20), pharmacists (N=20), and corporate leaders (N=20). Interviews will assess perceptions towards screening/intervention, internal organizational challenges, and processes related to ABI-MTM implementation for large-scale research and practice. Altogether, results of this study will provide critical insights, foundational data, and strategies for executing a powered trial and possible future system/practice-level implementation.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* ≥18 years
* Not receiving cancer treatment
* Current alcohol use
* Prescribed an opioid medication

Exclusion Criteria:

* SA 2 exclusion
* Are pregnant
* Cannot provide collateral contact information for ≥2 persons
* Do not have a reliable land line or mobile phone to be contacted by study staff
* Are filling only buprenorphine
* Plan to leave the area for an extended period of time in the next 3-months, or
* Have experienced a psychotic and/or manic episode in the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Cochran, Principal Investigator — University of Utah
Locations (1):
- University of Tennessee College of Medicine, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Qualitative Interviews: Interviews were conducted of pharmacy technicians, pharmacists, and corporate leaders. Interviews assessed perceptions towards screening/intervention, internal organizational challenges, and processes related to ABI-MTM implementation for large-scale research and practice.
Period: Overall Study
Arm/Group | Alcohol-targeted Brief Intervention-Medication Therapy Management | Standard Medication Counseling | Qualitative Interviews
Started | 22 | 22 | 68
Completed | 22 | 22 | 68
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol-targeted Brief Intervention-Medication Therapy Management | Standard Medication Counseling | Qualitative Interviews | Total
Number analyzed (Participants) | 22 | 22 | 68 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 10 | 68 | 92
  >=65 years | 8 | 12 | 0 | 20
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Males | 14 | 15 | 26 | 55
  Females | 8 | 17 | 36 | 61
  Unknown | 0 | 0 | 6 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 22 | 21 | 0 | 43
  Unknown or Not Reported | 0 | 0 | 68 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 20 | 22 | 0 | 42
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 68 | 68
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 68 | 112

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Use Reductions
Description: The investigators will use the Timeline Follow Back to assess alcohol use reductions. This measure is a calendar based assessment that captures a continuous number (counts) of days of substance use. This quantitative measure is both valid and reliable.
Time Frame: 3 Months. Changes in alcohol use will be assessed by comparing baseline to month 2. Changes in alcohol use will also be assessed by comparing month 2 to month 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol-targeted Brief Intervention-Medication Therapy Management | Standard Medication Counseling
Number analyzed (Participants) | 22 | 22
Participants
  <=19% reduction in drinks per day | 11 | 12
  20-24% reduction in drinks per day | 1 | 1
  25-29% reduction in drinks per day | 1 | 2
  >=30% reduction in drinks per day | 9 | 7

2. Primary Outcome: Opioid Medication Use
Description: The investigators will use the Treatment Services Review 6 to assess if the patients decrease their medication use. This measure is a calendar based assessment that captures a continuous number (counts) of days of substance use. This quantitative measure is both valid and reliable.
Time Frame: 3 Months. Changes in medication use will be assessed by comparing baseline to month 2. Changes in medication use will also be assessed by comparing month 2 to month 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Alcohol-targeted Brief Intervention-Medication Therapy Management | Standard Medication Counseling
Number analyzed (Participants) | 22 | 22
Participants
  <=10% reduction in morphine milligram equivalents | 12 | 17
  11-19% reduction in morphine milligram equivalents | 1 | 0
  20-24% reduction in morphine milligram equivalents | 1 | 0
  25-29% reduction in morphine milligram equivalents | 1 | 1
  >=30% reduction in morphine milligram equivalents | 7 | 4

ADVERSE EVENTS:
Time Frame: This was a minimal risk study and as such no adverse events were collected.
Description: All cause mortality, serious adverse events, and other (not including serious) adverse events were not monitored.
Arm/Group | Alcohol-targeted Brief Intervention-Medication Therapy Management | Standard Medication Counseling
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/72/NCT05599672/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT05599672/ICF_001.pdf